CLINICAL TRIAL: NCT04720001
Title: Florbetaben PET Imaging in Primary Progressive Aphasia
Brief Title: Florbetaben PET Imaging in PPA
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Collaborators: Northwestern University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB23-1360
Record Dates: First submitted 2021-01-19; First posted 2021-01-22 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2022-02

CONDITIONS: Primary Progressive Aphasia; Alzheimer Disease
Keywords: Alzheimer's Disease; Dementia; Primary Progressive Aphasia; Neurocognitive Disorders; Speech Disorders
MeSH Terms: conditions — Aphasia, Primary Progressive; Alzheimer Disease; Dementia; Neurocognitive Disorders; Speech Disorders | interventions — 4-(N-methylamino)-4'-(2-(2-(2-fluoroethoxy)ethoxy)ethoxy)stilbene

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Experimental: Florbetaben F18 recipients: Participants in this arm of the study will receive 8.1mCi of florbetaben F18 and then be scanned in a PET scanner for brain imaging.
  Interventions: Drug: Florbetaben F18; Device: PET

INTERVENTIONS:
Drug: Florbetaben F18 — A single injection of 8.1mCi of florbetaben F18 will be administered by intravenous bolus injection
  Other Names: trade name NeuraCeq
Device: PET — PET Scan for brain imaging

SUMMARY:
The purpose of this research is to better understand how dementia affects activity in different parts of the brain.

DETAILED DESCRIPTION:
This study will examine Positron Emission Tomography (PET) imaging with Florbetaben F18. Florbetaben F18 is a radioactive tracer that binds to particles in your brain. This process displays activity in the brain. Florbetaben F18 is a PET amyloid imaging agent approved by the United States Food and Drug Administration (FDA) to estimate the amount of beta-amyloid plaque in adult patients who are being evaluated for Alzheimer's disease and other causes of cognitive decline. The purpose of this research is to better understand how dementia affects activity in different parts of the brain. Currently, the scientific community is limited by how well it can see inside the brain. The use of a PET scan better helps us understand what the brain looks like in a diseased state. Participation in the study will help to understand what brain activity looks like, especially around language regions.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a diagnosis of PPA or a related dementia syndrome

Exclusion Criteria:

* Pregnant
* Breastfeeding
* Receiving radiation clinically

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from other research projects at Northwestern's Mesulam Center. Some of these projects recruit participants from the local Chicagoland area and others recruit participants from across the United States. As Primary Progressive Aphasia is an uncommon syndrome, participant recruitment is not focused on a specific demographic area.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2018-08-23 (Actual); Primary Completion 2021-01-21 (Actual); Study Completion 2021-02-26 (Actual)

PRIMARY OUTCOMES:
Amyloid plaque levels in PPA participants | 2 Years
  Amyloid plaque aggregation as measured by florbetaben F18 standard uptake value ratio cerebral and cerebellar regions of interest.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Rogalski, Ph.D, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago - American School Building, Chicago, Illinois, United States